CLINICAL TRIAL: NCT02331121
Title: Multimedia First Aid Program for Families
Acronym: FirstAid_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SBIR82RR-II; R43HD049156 (NIH)
Record Dates: First submitted 2014-06-21; First posted 2015-01-06 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Injury
Keywords: children; parents; internet; video; training; interactive
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text-only Online Training (Active Comparator): Text-only evidence-based training content on CPR, choking relief & first aid
  Interventions: Behavioral: Text-only Online Training
- Family First Aid Online Training (Experimental): Interactive multimedia evidence-based training content on CPR, choking relief & first aid
  Interventions: Behavioral: Family First Aid Online Training

INTERVENTIONS:
Behavioral: Family First Aid Online Training — Web-based interactive multimedia program comprised of videos, interactive animations and text information designed to teach parents of children aged birth to 12 years old basic first-aid and CPR skills, including the option to practice skills as needed.
  Arms: Family First Aid Online Training
Behavioral: Text-only Online Training — Online text created from the American Heart Association's 2010 guidelines for CPR training via a computer, depicting infant, child and adult CPR skills and choking relief.
  Arms: Text-only Online Training

SUMMARY:
Unintentional injuries are the leading cause of death for children and infants under 14 years of age. Many of these deaths are preventable, in part by promoting injury prevention behaviors but also by administering effective emergency first aid techniques until advanced care arrives. This project created a web site program that paired video-based instruction with interactive skills training to teach parents of children birth to 12 years old basic first-aid and CPR skills, and that included the option to practice skills as needed.

DETAILED DESCRIPTION:
Program content was based on the American Heart Association's (AHA) 2010 guidelines for CPR and first aid training. The Online IMM course was designed to teach participants in six modules: Principles of care; CPR for infants; CPR for children; How to relieve infant choking; How to relieve child choking; and Preventing injuries. Participants were also able to view text articles on first aid topics, such as Wound care or Caring for burns. Although the users of the Online IMM training program did not have direct contact with a manikin during their training, there were opportunities to practice CPR skills through the use of interactive animations. These animations demonstrated and then encouraged users to practice key functions similar to actual CPR skill delivery: including the location, depth and rate of compressions, opening the airway and giving breaths. Participants were encouraged to view the entire program; however, they could navigate and review all program content as much or as little as desired.

ELIGIBILITY:
Inclusion Criteria:

* Parents or guardians of children aged newborn to 12 years old could potentially be as young as 18 years old. Parents or legal guardians could potentially be as old as 65 or older.
* Children under the age of 18 were not included, even with parental consent, because of the online nature of the study and inability to verify parental consoent.

Exclusion Criteria:

* Only English-speaking participants were accepted because the program was developed only for English speakers.
* All English-speaking parents of children aged newborn - 12 years old who wished to participate were included.
* There were no exclusions based on race/ethnicity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Knowledge (knowledge score was calculated by summing the number of items answered correctly and dividing by the total number of items to arrive at the percent of items correctly endorsed.) | 40-day follow-up
  A knowledge score was calculated by summing the number of items answered correctly and dividing by the total number of items to arrive at the percent of items correctly endorsed.

SECONDARY OUTCOMES:
Self-efficacy (assessed with a 5-point scale) | 10-day posttest and 40-day follow-up
  Change in self-efficacy to perform CPR and choking relief skills was assessed with a 27- item scale (e.g., How confident are you that you know the correct ratio of compressions to breaths for CPR for a younger child ages 1-8) assessed with a 5-point scale (1=not at all confident; 5=extremely confident; alpha = .97).

CONTACTS AND LOCATIONS:
Overall Officials: Amelia J Birney, MPH, MCHES, Principal Investigator — Oregon Center for Applied Science
Locations (1):
- Oregon Center for Applied Science, Eugene, Oregon, United States